CLINICAL TRIAL: NCT03709875
Title: A Cost-effective Analysis of Telerehabilitation in Patients With Severe Acquired Brain Injury
Brief Title: Telerehabilitation in Severe Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Collaborators: IRCCS San Camillo, Venezia, Italy (Other); University of Messina (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Professor, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/2018
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Brain Injuries; Stroke
Keywords: Telerehabilitation; Motor outcomes; Cognitive dysfunction
MeSH Terms: conditions — Brain Injuries; Stroke; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: multi-center, prospective, parallel design, single-blind trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TR Treatment (Experimental): TR will be delivered by means of an advanced video-conferencing system, and patients will be provided with low-cost monitoring devices, able to collect data about the health status and QoL. All treatments from remote are based on scheduled videoconferences between the patient's home and the Clinical Units, and therapists can control and modify the exercises. A virtual reality based system, consisting of two PC-based workstations, located at the patient's home and at the rehabilitation center, will be used. For the motor treatments the patient has to move the real end effector, following the trajectory of the corresponding virtual task displayed on his computer screen. The speech and cognitive exercises will be delivered from the two Research Institutes to the patient's home.
  Interventions: Device: TR Treatment
- Conventional Treatment (Other): In this group patients will be treated with conventional physiotherapy and speech training, adjusted in reason of the clinical needs, as usually. Treatments for motor limbs activity will be focused on functional active-assistive and active exercises. Conventional "paper and pencil" training will be used to improve cognitive function.
  Interventions: Device: TR Treatment

INTERVENTIONS:
Device: TR Treatment — A virtual reality based system, consisting of two PC-based workstations, located at the patient's home and at the rehabilitation center, will be used. For the motor treatments the patient has to move the real end effector, following the trajectory of the corresponding virtual task displayed on his computer screen. The speech (mainly lexical based) and cognitive (attention focused) exercises will be delivered from the two Research Institutes to the patient's home. During the treatment at home, the patients will use wearable monitoring devices to monitor their status (speed, heart rate, respiratory rate, training load and single-lead ECG in real-time) and to provide real-time feedback during exercises.

SUMMARY:
We will investigate the use of TR, based on advanced Information and Communication Technology (ICT) solutions, taking into account that the supervision of rehabilitation at home will be enriched with the counselling and vital parameters monitoring. The aim of the study is to evaluate that TR is at least non-inferior in comparison with the same amount of usual territorial rehabilitative physical treatments (UTRT), taking into account patients' functional recovery, psychological well-being, caregiver burden, and healthcare costs. The enrolled patients will be balanced for pathology and randomized in two groups, performing TR (G1) or standard rehabilitation training (G2), respectively, according to a pc-generated random assignment.TR will be delivered by means of an advanced video-conferencing system, whereas the patient will be provided with low-cost monitoring devices, able to collect data about his/her health status and QoL. In both the groups each treatment (either cognitive or motor, or both as per patient functional status) will last about one hour a day, five days/week, for 12 weeks. Two structured telephone interviews will be administered to the patients (when possible) and/or their caregivers, and to all the healthcare professionals involved in the patient management, one week after the beginning and at the end of the TR.

ELIGIBILITY:
Inclusion Criteria:age range 18 to 65 years; diagnosis of SABI; availability at home internet connection.

Exclusion Criteria: severe cognitive and behavioral impairments, cardio-respiratory instability or other medical illness potentially interfering with the treatment, severe limb spasticity, high-risk of spontaneous fracture, substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-26 (Estimated); Primary Completion 2019-05-27 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
WHO Disability Assessment schedule | 3 months
  This generic assessment instrument for health and disability may be considered a tool to produce standardized disability levels and profiles. It is applicable across cultures, in all adult populations, and is directly linked at the level of the concepts to the International Classification of Functioning, Disability and Health (ICF).
Montreal Cognitive assessment | 3 months
  he Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.he MoCA test is a one-page 30-point test administered in approximately 10 minutes.

SECONDARY OUTCOMES:
Fugl- Meyer for Upper limb | 3 months
  The Fugl-Meyer Upper Extremity (FMUE) Scale1 is a widely used and highly recommended stroke-specific, performance-based measure of impairment. It is designed to assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. It has been extensively used as an outcome measure in rehabilitation trials and to record post-stroke recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco S Calabrò, PhD, Principal Investigator — IRCCS Centro Neurolesi
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calabro RS, Bonanno M, Torregrossa W, Cacciante L, Celesti A, Rifici C, Tonin P, De Luca R, Quartarone A. Benefits of Telerehabilitation for Patients With Severe Acquired Brain Injury: Promising Results From a Multicenter Randomized Controlled Trial Using Nonimmersive Virtual Reality. J Med Internet Res. 2023 Aug 21;25:e45458. doi: 10.2196/45458. PMID 37490017